CLINICAL TRIAL: NCT05749926
Title: Immunogenicity and Reactogenicity of the Beta-variant Recombinant Protein Booster Vaccine (VidPrevtyn Beta, Sanofi) Compared to a Bivalent mRNA Vaccine (Comirnaty Original/Omicron BA.4-5, BioNTech-Pfizer) in Adults Previously Vaccinated With at Least 3 Doses of COVID-19 mRNA Vaccine: A Non-inferiority Multicenter Single-blinded, Randomized Trial
Brief Title: Immunogenicity and Reactogenicity of the Beta-variant Recombinant Protein Booster Vaccine (VidPrevtyn Beta, Sanofi) Compared to a Bivalent mRNA Vaccine (Comirnaty Original/Omicron BA.4-5, BioNTech-Pfizer) in Adults Previously Vaccinated With at Least 3 Doses of COVID-19 mRNA Vaccine
Acronym: CoviBOOST 2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: IREIVAC/COVIREIVAC Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APHP220775; 2022-002715-38 (EudraCT Number)
Record Dates: First submitted 2023-02-28; First posted 2023-03-01 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Vaccine Reaction; COVID-19
Keywords: COVID 19; mRNA vaccines; Immunulogy; Sub-unit vaccine; Booster
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comirnaty® BNT162b2 /Omicron BA.4-5 vaccine (Pfizer-BioNTech) (Active Comparator): Length of use : 1 day
  Interventions: Biological: Comirnaty® BNT162b2 /Omicron BA.4-5 vaccine (Pfizer-BioNTech)
- VidPrevtyn® Beta vaccine (Sanofi/GSK) (Experimental): Length of use : 1 day
  Interventions: Biological: VidPrevtyn® Beta vaccine (Sanofi/GSK)

INTERVENTIONS:
Biological: Comirnaty® BNT162b2 /Omicron BA.4-5 vaccine (Pfizer-BioNTech) — A single administration of COVID-19 vaccine will be performed at D0, depending on randomization
  Arms: Comirnaty® BNT162b2 /Omicron BA.4-5 vaccine (Pfizer-BioNTech)
Biological: VidPrevtyn® Beta vaccine (Sanofi/GSK) — A single administration of COVID-19 vaccine will be performed at D0, depending on randomization
  Arms: VidPrevtyn® Beta vaccine (Sanofi/GSK)

SUMMARY:
The objective of this trial is to compare the immunogenicity and the safety of the Beta-variant recombinant protein booster vaccine (VidPrevtyn® Beta, Sanofi) to a bivalent mRNA vaccine (Comirnaty Original/Omicron BA.4-5, BioNTech-Pfizer) in adults previously vaccinated with at least 3 doses of COVID-19 mRNA vaccine. The results will provide important data for the future COVID 19 vaccine strategy.

A biobank will also be set up to evaluate the protection conferred by one or other of these vaccines as booster in the event of the emergence of new variants in the future.

DETAILED DESCRIPTION:
The efficacy of COVID 19 vaccines for reducing the risk of severe COVID-19 infection is demonstrated in real life.

However, data currently available on the persistence of immunity after vaccination on the one hand and the emergence of viral variants with reduced sensibility to vaccine immunity on the other, raise the need to administer boosters to maintain the protection and to compare different strategies as bivalent mRNA vaccines but also others platforms.

The vaccines currently recommended as boosters in France are mRNA bivalent vaccines, adapted to better match the circulating variants of SARS-CoV-2 and expected to provide broader protection against Omicron sub variants (19). However, the rapid antigenic evolution of SARS-CoV-2 and the antigenic imprinting against the initial Hu-1 strain could reduce their effectiveness.

More recently, the Beta-variant recombinant protein booster vaccine (VidPrevtyn Beta, Sanofi) obtained European authorization and is recommended in France as booster as an alternative to the bivalent mRNA vaccines (21, 22). However, in the absence of comparative data with the bivalent mRNA vaccines, VidPrevtyn Beta is recommended as second line.

It has been shown with vectored vaccines that a heterologous vaccination scheme could be more immunogenic than a homologous scheme (23). Our group previously showed that VidPrevtyn Beta, administered as a third vaccine dose, induces higher immune response than the mRNA BNT162b2 vaccine (Comirnaty, BioNTech-Pfizer), against Beta variant but also others variants of concern (VOC) including Omicron BA1 (20) and Omicron BA4/5 (data submitted for publication). The data available at 3 and 6 months after the boost, show that VidPrevtyn Beta could be also of interest in term of durability of the response (data not published). The hypothesis is that a Beta variant protein recombinant vaccine could enlarge the protection against the variants by overpassing antigenic imprinting and the adjuvant improve the duration of immune response and protection. Moreover, the Beta-variant recombinant protein vaccine could bring an advantage in terms of reactogenicity, acceptability, cost and accessibility.

In this context, as recently pointed by the HAS, comparative data on immunogenicity and reactogenicity between a bivalent mRNA vaccine and the Beta-variant recombinant protein, both administered as boosters, are needed to better adapt the COVID 19 vaccine recommendations for the future.

This study is Comparative, non-inferiority, single-blinded, multicenter, randomized trial.

Randomization in a 1:1 ratio, will be stratified by age (18-60 years and ≥ 60 years of age) and history of SARS-CoV-2 infection

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years and over
2. Adult in a healthy condition or with a stable health status, determined by medical history, targeted physical examination and clinical judgement of the investigator to be in stable state of health. Participants with pre-existing stable chronic medical conditions defined as condition not requiring significant change in therapy or hospitalization for worsening disease within 4 weeks from enrollment can be included at the discretion of the investigator.
3. For women of childbearing age: a negative highly sensitive pregnancy urinary test during the inclusion visit
4. Confirmed receipt of at least three doses of COVID-19 mRNA vaccine the last dose at least 6 months prior to study vaccine
5. Understands and agrees to comply with the study procedures
6. Written informed consent signed by both the participant and the investigator
7. Subject affiliated to the French Social Security System.

Exclusion Criteria:

1. Acute febrile infection (body temperature ≥ 38.0°C) within the previous 72 hours and/or presenting symptoms suggestive of COVID-19 within the previous 28 days
2. Confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection < 3 months prior to the study vaccine dose.
3. Immunosuppressive therapy such as corticosteroids > 10 mg prednisone equivalent/day (excluding topical preparations and inhalers) within 3 months prior to inclusion or within 6 months for chemotherapies.
4. Treatment with immunoglobulins or other blood derivatives within 3 months prior to inclusion or scheduled administration of immunoglobulins or blood derivatives before the end of the study.
5. Any medical condition, such as cancer, that might impair the immune response.
6. Use of experimental immunoglobulins, experimental monoclonal antibodies or convalescent plasma is not permitted during the study.
7. Pregnancy or breastfeeding currently ongoing
8. History of severe adverse events following vaccine administration including anaphylactic reaction and associated symptoms such as rash, breathing problems, angioedema, and abdominal pain, or a history of allergic reaction that could be triggered by a component of the SARS-COV-2 vaccine at the time of the first vaccine injection:
9. Any bleeding disorder considered as a contraindication to an intramuscular injection,
10. Participation in other interventional research involving humans within 4 weeks prior to the inclusion visit, or participation in any other vaccine trial excepted for those with mid or long term follow up when vaccination was made at least 4 weeks before the injection in the study. In this case no delay is required after the end of the study participation".
11. Subject under legal protection (e.g. guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2023-05-16 (Actual); Primary Completion 2023-07-12 (Estimated); Study Completion 2024-07-12 (Estimated)

PRIMARY OUTCOMES:
Neutralizing antibody titers against the SARS-CoV-2 variant of most prominent public health interest and against one of the variant targeted by the vaccines | 28 Days
  Title : Neutralizing antibody titers against the SARS-CoV-2 variant of most prominent public health interest and against one of the variant targeted by the vaccines Time Frame : 28 Days
  Description:
  There will be a coprimary endpoint : Neutralizing antibody titers against the SARS-CoV-2 variant of most prominent public health interest according to pandemic evolution (among D614G, B.1.351, Omicron sub-variants BA.4-5, BQ1.1 and XBB or another recent variant) and against one of the variant targeted by the vaccines. The two variants will be specified in the statistical analysis plan before D28 data base lock.
  Neutralizing antibody titers will be measured by a microneutralization technique 28 days after the booster dose.

SECONDARY OUTCOMES:
Humoral immune response against SARS-CoV-2 variants | Day0, Day15, Day28, 3 Months, 6 Months and 12 Months
  1. Neutralizing antibody titers
     1. Neutralizing antibody titers against SARS-CoV-2 D614G, and variants B.1.351, Omicron sub-variants BA.4-5, BQ1.1 and XBB (or another recent variant of prominent public health interest according to pandemic evolution), measured by a microneutralization technique.
     2. Seroresponse rate in each group. Seroresponse is defined as a 10 fold or greater rise in serum neutralization titer at each follow-up time relative to D0.
  2. ELISA:
     Anti-Spike IgG levels expressed as BAU/mL, according to WHO recommendations.
  3. LUMINEX:
     1. Antibodies to CTD domain of the SARS-CoV-2 N protein to detect recent natural infections.
     2. Full length Spike protein expressed as BAU/mL)
     3. Antibodies to RBD of Wuhan, B.1.1.7, B.1.617.2, B.1.351, Omicron BA.1/2/5, BQ1.1, XBB and others variants according to pandemic evolution.
Number and intensity of local and systemic adverse | 7 and 28 days
  Number and intensity of local and systemic adverse events of any degree occurring up to day 7 after administration of the booster dose (assessed from the list of solicited adverse events); number and intensity of unsolicited clinical events up to 28 days
Factors of interest | Day 0
  Factors of interest are age, gender, previous SARS-COV-2 infection, time interval between the last dose of vaccine and the booster dose, and vaccine boost type
Cellular immune response | Day 0, Day 7, Day 15, Month 3
  1. ELISpot IFN-IL-2 CD4 and CD8 response at D0 and D15 (ancillary study) against B1.351, BA.5, BQ1.1, XBB.1 ;
  2. Repertoire analysis of Memory Spike specific B cells and early ASC response at D0, D7 and M3.
Number of Covid 19 cases | Day 7 up to Month 12
  Number of Covid 19 cases (symptomatic with PCR or Ag positive tests, or asymptomatic with anti NP antibodies increase from D7 to M12)

CONTACTS AND LOCATIONS:
Locations (1):
- CIC 1417 Cochin-Pasteur, Paris, France

IPD SHARING:
Plan to Share IPD: No
The IPD will not be share. The 2 vaccines used in this study are marketed vaccine and used in routine care.